CLINICAL TRIAL: NCT00561158
Title: Dietary Changes in African American Women By Activation
Brief Title: Eat Well Live Well Nutrition Program
Acronym: EWLW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: St. Louis University (Other); Grace Hill Health Centers, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK48134 (completed); R01DK048143 (NIH)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes or Diabetes Prevention
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Behavioral: Eat Well Live Well Nutrition Program
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Eat Well Live Well Nutrition Program — 12 sessions (6 group and 6 individual)over a period of 3 months with a 3 month follow-up period. The group sessions involve active learning exercises crucial to learning and utilizing nutrition information.
  The group sessions included are:
  * Rate Your Plate: determining high fat foods
  * Label Reading: reading food labels
  * Comparison Shopping: using unit pricing labels maximize nutritional value on a limited income
  * Recipe Modification: preparing old recipes in new ways to reduce fat
  * Eating Out: order healthier fast foods
  * Coping with High Risk Situations: coping with situations in which these new habits may be threatened
  Six individual sessions will introduce participants to low fat eating patterns or ways to lower fat in their diet, including:
  * Substituting fat-modified foods for high fat foods
  * Avoiding fat as a seasoning or flavoring
  * Avoiding fried foods
  * Modifying meat
  * Replacing high fat foods with fruits, vegetables, grains and breads
  Arms: A

SUMMARY:
The purpose of the study is to develop and evaluate a dietary change program specifically for low-income, African-American women who are at risk for developing diabetes due to obesity. The program uses an innovative approach that emphasizes risk awareness, self-efficacy, and skills training through active learning exercises related to healthy eating. The program is delivered by peer educators in the community and addresses economic and cultural factors that are very important to program participants.

ELIGIBILITY:
Inclusion Criteria:

* African-American Women
* Aged 25-55 years
* No current diabetes, obese (20% over ideal body weight)
* In community neighborhoods

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 398 (Actual)
Dates: Start 1994-06; Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Weight & Body Mass Index (BMI) | pre-, post and three month follow-up
Fat intake (measured by Food Frequency Questionnaire) including: percent calories from fat, percent calories from saturated fat.

SECONDARY OUTCOMES:
Depressive symptoms (C-ESD) | pre-, post and three month follow-up
Dietary Knowledge: ten items that test knowledge of: i) fat in foods that are specific to target population; ii) Label Reading; iii) modifying recipes to lower fat content; and iv) saturated versus unsaturated fats | pre-, post and three month follow-up
Eating Habits: assessed using Eating Patterns Questionnaire, a 1993 revised version of Food Habits Questionnaire developed by Kristal, Shattuck & Henry | pre-, post and three month follow-up
Attitudes about fat in diet
Cultural relevancy

CONTACTS AND LOCATIONS:
Overall Officials: Wendy F Auslander, PhD, Principal Investigator — Washington University School of Medicine